CLINICAL TRIAL: NCT03104400
Title: A Phase 3, Randomized, Double-Blind, Study Comparing Upadacitinib (ABT-494) to Placebo and to Adalimumab in Subjects With Active Psoriatic Arthritis Who Have a History of Inadequate Response to at Least One Non-Biologic Disease Modifying Anti-Rheumatic Drug (DMARD) - SELECT - PsA 1
Brief Title: A Study Comparing Upadacitinib (ABT-494) to Placebo and to Adalimumab in Participants With Psoriatic Arthritis Who Have an Inadequate Response to at Least One Non-Biologic Disease Modifying Anti-Rheumatic Drug (DMARD)
Acronym: SELECT - PsA 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-572; 2016-004130-24 (EudraCT Number)
Record Dates: First submitted 2017-04-04; First posted 2017-04-07 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Psoriatic Arthritis
Keywords: Arthritis; Psoriasis; Anti-inflammatory; Joint disease; Musculoskeletal disease; Anti-Rheumatic
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis; Psoriasis; Joint Diseases; Musculoskeletal Diseases | interventions — Adalimumab; upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Upadacitinib 15 mg (Experimental): Period 1: Participants receive upadacitinib 15 mg orally once a day (QD) and matching placebo to adalimumab by subcutaneous injection every other week (EOW) for 56 weeks.
  Period 2: Participants will continue to receive upadacitinib 15 mg once daily.
  Interventions: Drug: Upadacitinib; Drug: Placebo to Adalimumab
- Upadacitinib 30 mg (Experimental): Period 1: Participants receive upadacitinib 30 mg orally once a day and matching placebo to adalimumab by subcutaneous injection every other week for 56 weeks.
  Period 2: Participants will continue to receive upadacitinib 30 mg once daily.
  Interventions: Drug: Upadacitinib; Drug: Placebo to Adalimumab
- Adalimumab (Active Comparator): Period 1: Participants receive adalimumab 40 mg by subcutaneous injection every other week and matching placebo to upadacitinib orally QD for 56 weeks.
  Period 2: Participants continue to receive adalimumab 40 mg every other week.
  Interventions: Drug: Adalimumab; Drug: Placebo to Upadacitinib
- Placebo / Upadacitinib 15 mg (Placebo Comparator): Period 1: Participants receive matching placebo to upadacitinib orally once a day for 24 weeks then upadacitinib 15 mg once daily for 32 weeks, and matching placebo to adalimumab by subcutaneous injection EOW for the entire 56 weeks.
  Period 2: Participants will continue to receive upadacitinib 15 mg once daily.
  Interventions: Drug: Upadacitinib; Drug: Placebo to Upadacitinib; Drug: Placebo to Adalimumab
- Placebo / Upadacitinib 30 mg (Placebo Comparator): Period 1: Participants receive matching placebo to upadacitinib orally once a day for 24 weeks then upadacitinib 30 mg once daily for 32 weeks, and matching placebo to adalimumab by subcutaneous injection EOW for the entire 56 weeks.
  Period 2: Participants will continue to receive upadacitinib 30 mg once daily.
  Interventions: Drug: Upadacitinib; Drug: Placebo to Upadacitinib; Drug: Placebo to Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Administered by subcutaneous injection
  Other Names: Humira®
  Arms: Adalimumab
Drug: Upadacitinib — Oral tablet
  Other Names: ABT 494; RINVOQ®
  Arms: Placebo / Upadacitinib 15 mg; Placebo / Upadacitinib 30 mg; Upadacitinib 15 mg; Upadacitinib 30 mg
Drug: Placebo to Upadacitinib — Oral tablet
  Arms: Adalimumab; Placebo / Upadacitinib 15 mg; Placebo / Upadacitinib 30 mg
Drug: Placebo to Adalimumab — Administered by subcutaneous injection
  Arms: Placebo / Upadacitinib 15 mg; Placebo / Upadacitinib 30 mg; Upadacitinib 15 mg; Upadacitinib 30 mg

SUMMARY:
This study includes two periods. The main objective of Period 1 is to compare the efficacy of upadacitinib 15 mg once daily (QD) and 30 mg QD versus placebo and versus adalimumab (Humira®) in participants with moderately to severely active psoriatic arthritis (PsA) who have had an inadequate response to non-biologic DMARDs (DMARD-IR). Period 1 is also designed to compare the efficacy of upadacitinib 15 mg and 30 mg QD versus placebo for the prevention of structural progression.

The objective of Period 2 is to evaluate the long-term safety, tolerability and efficacy of upadacitinib 15 mg and 30 mg QD in participants who have completed Period 1.

DETAILED DESCRIPTION:
The study includes a 35-day screening period, a 56-week blinded period (Period 1), a long-term extension period of up to a total treatment duration of approximately 5 years (Period 2), a 30-day follow-up call or visit, and a 70-day follow-up call.

Period 1 includes 24 weeks of randomized, double-blind, placebo-controlled and active comparator-controlled treatment followed by 32 weeks of active comparator-controlled upadacitinib; at Week 24 participants assigned to placebo will be switched to upadacitinib according to their randomization assignment.

Participants who meet eligibility criteria will be randomized in a 2:2:2:1:1 ratio to one of five treatment groups:

* Group 1: Upadacitinib 15 mg QD
* Group 2: Upadacitinib 30 mg QD
* Group 3: Adalimumab 40 mg every other week (EOW)
* Group 4: Placebo followed by upadacitinib 15 mg QD
* Group 5: Placebo followed by upadacitinib 30 mg QD

Randomization will be stratified by extent of psoriasis (≥ 3% body surface area [BSA] or < 3% BSA), current use of at least 1 non-biologic DMARD, presence of dactylitis, and presence of enthesitis, except for participants from China and Japan, where randomization for each country will be stratified by extent of psoriasis (≥ 3% BSA or < 3% BSA) only.

Participants who complete the Week 56 visit (end of Period 1) will enter the long-term extension portion of the study, Period 2 (total treatment up to approximately 5 years), and continue study treatment as assigned in Period 1 in a blinded manner until the last subject completes the last visit of Period 1 (Week 56), when study drug assignment in both periods will be unblinded and participants will be dispensed study drug in an open-label fashion until the completion of Period 2.

At Week 16, rescue therapy will be offered to participants classified as non-responders (defined as not achieving at least 20% improvement in tender joint count (TJC) and / or swollen joint count (SJC) at both Week 12 and Week 16). Starting at Week 36, participants who fail to demonstrate at least 20% improvement in either or both TJC and SJC compared to Baseline at 2 consecutive visits will be discontinued from study drug treatment. Additionally, in participants continuing on study drug, starting at the Week 36 visit, initiation of or change in background PsA medication(s) is allowed as per local label.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PsA with symptom onset at least 6 months prior to the Screening Visit and fulfillment of the Classification Criteria for PsA (CASPAR) criteria.
* Participant has active disease at Baseline defined as >= 3 tender joints (based on 68 joint counts) and >= 3 swollen joints (based on 66 joint counts) at Screening and Baseline Visits.
* Presence of either at Screening:

  1. >= 1 erosion on x-ray as determined by central imaging review or;
  2. high-sensitivity C-reactive protein (hs-CRP) > laboratory defined upper limit of normal (ULN).
* Diagnosis of active plaque psoriasis or documented history of plaque psoriasis.
* Participant has had an inadequate response (lack of efficacy after a minimum 12 week duration of therapy) to previous or current treatment with at least 1 non-biologic DMARD at maximally tolerated dose (methotrexate (MTX), sulfasalazine (SSZ), leflunomide (LEF), cyclosporine, apremilast, bucillamin or iguratimod), or participant has an intolerance to or contraindication for DMARDs as defined by the investigator.
* Participant who is on current treatment with concomitant non-biologic DMARDs at study entry must be on <= 2 non-biologic DMARDs (except the combination of MTX and leflunomide). The following non-biologic DMARDs are allowed: MTX, sulfasalazine, leflunomide, apremilast, hydroxychloroquine (HCQ) , bucillamine or iguratimod, and have been ongoing for >= 12 weeks and at stable dose for >= 4 weeks prior to the Baseline Visit. No other DMARDs are permitted during the study.

  i. Participants who need to discontinue DMARDs prior to the Baseline Visit to comply with this inclusion criterion must follow the procedure specified below or at least five times the mean terminal elimination half-life of a drug:
  1. >= 8 weeks for LEF if no elimination procedure was followed, or adhere to an elimination procedure (i.e., 11 days with cholestyramine, or 30 days washout with activated charcoal or as per local label);
  2. >= 4 weeks for all others.

     Exclusion Criteria:
* Prior exposure to any Janus Kinase (JAK) inhibitor (including but not limited to ruxolitinib, tofacitinib, baricitinib, and filgotinib).
* Current treatment with > 2 non-biologic DMARDs; or use of DMARDs other than methotrexate, sulfasalazine, leflunomide, apremilast, hydroxychloroquine, bucillamine, or iguratimod; or use of methotrexate in combination with leflunomide.
* History of fibromyalgia, any arthritis with onset prior to age 17 years, or current diagnosis of inflammatory joint disease other than PsA (including, but not limited to rheumatoid arthritis, gout, overlap connective tissue diseases, scleroderma, polymyositis, dermatomyositis, systemic lupus erythematosus). Prior history of reactive arthritis or axial spondyloarthritis including ankylosing spondylitis and nonradiographic axial spondyloarthritis is permitted if documentation of change in diagnosis to PsA or additional diagnosis of PsA is made. Prior history of fibromyalgia is permitted if documentation of change in diagnosis to PsA or documentation that the diagnosis of fibromyalgia was made incorrectly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1705 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (345):
- United States (114):
  - Rheum Assoc of North Alabama /ID# 163231, Huntsville, Alabama
  - SunValley Arthritis Center, Lt /ID# 161221, Peoria, Arizona
  - AZ Arthritis and Rheumotology Research, PLLC /ID# 159981, Phoenix, Arizona
  - AZ Arthritis and Rheumotology Research, PLLC /ID# 160033, Phoenix, Arizona
  - AZ Arthritis and Rheumotology Research, PLLC /ID# 160036, Phoenix, Arizona
  - AZ Arthritis & Rheuma Research /ID# 160037, Phoenix, Arizona
  - AZ Arth & Rheum Res /ID# 166381, Tucson, Arizona
  - Little Rock Diagnostics Clinic /ID# 165161, Little Rock, Arkansas
  - Covina Arthritis Clinic /ID# 159891, Covina, California
  - St. Joseph Heritage Healthcare /ID# 159980, Fullerton, California
  - C.V. Mehta MD, Med Corporation /ID# 161216, Hemet, California
  - Care Access Research, Huntingt /ID# 160038, Huntington Beach, California
  - Kotha and Kotha /ID# 159823, La Mesa, California
  - TriWest Research Associates- La Mesa /ID# 159887, La Mesa, California
  - Arthritis & Osteo Medical Ctr /ID# 166760, La Palma, California
  - University of California, Los Angeles /ID# 164542, Los Angeles, California
  - VA Sacramento Medical Center /ID# 164196, Mather, California
  - East Bay Rheumatology Medical /ID# 166382, San Leandro, California
  - Inland Rheum Clin Trials Inc. /ID# 159828, Upland, California
  - Medvin Clinical Research /ID# 160034, Whittier, California
  - Denver Arthritis Clinic /ID# 159873, Denver, Colorado
  - Arthritis and Rheum Clin N. CO /ID# 160039, Fort Collins, Colorado
  - Colorado Arthritis Associates /ID# 159847, Lakewood, Colorado
  - Stamford Therapeutics Consorti /ID# 165131, Stamford, Connecticut
  - Clinical Res of West FL, Inc. /ID# 159829, Clearwater, Florida
  - International Medical Research - Daytona /ID# 160040, Daytona Beach, Florida
  - Omega Research Maitland, LLC /ID# 164193, DeBary, Florida
  - LeJenue Research Associates /ID# 170965, Miami, Florida
  - Precision Research Org, LLC /ID# 161287, Miami Lakes, Florida
  - Medallion Clinical Research Institute, LLC /ID# 161228, Naples, Florida
  - Millennium Research /ID# 159822, Ormond Beach, Florida
  - Arthritis Center, Inc. /ID# 163465, Palm Harbor, Florida
  - Gulf Region Clinical Res Inst /ID# 159851, Pensacola, Florida
  - BayCare Medical Group /ID# 159792, St. Petersburg, Florida
  - W. Broward Rheum Assoc Inc. /ID# 161388, Tamarac, Florida
  - Clinical Research of West Florida, Inc /ID# 160063, Tampa, Florida
  - University of South Florida /ID# 161286, Tampa, Florida
  - BayCare Medical Group, Inc. /ID# 159879, Tampa, Florida
  - Florida Medical Clinic /ID# 159992, Zephyrhills, Florida
  - Institute of Arthritis Researc /ID# 165873, Idaho Falls, Idaho
  - Advanced Clinical Research /ID# 159894, Meridian, Idaho
  - Great Lakes Clinical Trials /ID# 163435, Chicago, Illinois
  - OrthoIllinois /ID# 164546, Rockford, Illinois
  - Clinical Investigation Specialists - Skokie /ID# 160062, Skokie, Illinois
  - Deerbrook Medical Associates /ID# 159804, Vernon Hills, Illinois
  - Graves Gilbert Clinic /ID# 161285, Bowling Green, Kentucky
  - Four Rivers Clinical Research /ID# 159982, Paducah, Kentucky
  - Ochsner Clinic Foundation-New Orleans /ID# 165672, New Orleans, Louisiana
  - Johns Hopkins University /ID# 167665, Baltimore, Maryland
  - Klein & Associates, M.D., P.A. /ID# 164013, Cumberland, Maryland
  - The Center for Rheumatology & Bone Research /ID# 159874, Wheaton, Maryland
  - Tufts Medical Center /ID# 165144, Boston, Massachusetts
  - Mansfield Health Center /ID# 159805, Mansfield, Massachusetts
  - Clinical Pharmacology Study Gr /ID# 158700, Worcester, Massachusetts
  - Univ of Michigan Hospitals /ID# 164014, Ann Arbor, Michigan
  - Aa Mrc Llc /Id# 159846, Grand Blanc, Michigan
  - Advanced Rheumatology, PC /ID# 159893, Lansing, Michigan
  - Beals Institute PC /ID# 163128, Lansing, Michigan
  - Shores Rheumatology, PC /ID# 159889, Saint Clair Shores, Michigan
  - St. Luke's Hospital of Duluth /ID# 165671, Duluth, Minnesota
  - Clinvest Research LLC /ID# 161227, Springfield, Missouri
  - Clayton Medical Associates dba Saint Louis Rheumatology /ID# 159878, St Louis, Missouri
  - Glacier View Research Institut /ID# 167023, Kalispell, Montana
  - Westroads Clinical Research /ID# 159979, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center /ID# 161235, Lebanon, New Hampshire
  - Arthritis and Osteoporosis Associates /ID# 159802, Freehold, New Jersey
  - Atlantic Coast Research /ID# 159799, Toms River, New Jersey
  - Ocean Rheumatology, PA /ID# 163898, Toms River, New Jersey
  - Arthritis and Osteo Assoc /ID# 159994, Las Cruces, New Mexico
  - Santa Fe Rheumatology /ID# 163783, Santa Fe, New Mexico
  - NYU Langone Rheum Assoc /ID# 159985, Lake Success, New York
  - NYU Langone Medical Center /ID# 163230, New York, New York
  - St. Lawrence Health System /ID# 159848, Potsdam, New York
  - American Health Research /ID# 164354, Charlotte, North Carolina
  - DJL Clinical Research, PLLC /ID# 161390, Charlotte, North Carolina
  - M3-Emerging Medical Research, LLC /ID# 161391, Durham, North Carolina
  - Physicians East, PA /ID# 159872, Greenville, North Carolina
  - Cape Fear Arthritis Care /ID# 161224, Leland, North Carolina
  - Shanahan Rheuma & Immuno /ID# 159987, Raleigh, North Carolina
  - Trinity Health Med Arts Clinic /ID# 159800, Minot, North Dakota
  - MetroHealth Medical Center /ID# 159888, Cleveland, Ohio
  - The Ohio State University /ID# 159892, Columbus, Ohio
  - Clinical Research Source, Inc. /ID# 164545, Perrysburg, Ohio
  - STAT Research, Inc. /ID# 161392, Vandalia, Ohio
  - Health Research of Oklahoma /ID# 159880, Oklahoma City, Oklahoma
  - Altoona Ctr Clinical Res /ID# 159852, Duncansville, Pennsylvania
  - PA Regional Center /ID# 165670, Wyomissing, Pennsylvania
  - Articularis Healthcare Group, Inc d/b/a Low Country Rheumatology /ID# 163464, Summerville, South Carolina
  - West Tennessee Research Inst /ID# 159871, Jackson, Tennessee
  - Rheumatology Consultants, PLLC /ID# 159796, Knoxville, Tennessee
  - Dr. Ramesh Gupta /ID# 160061, Memphis, Tennessee
  - Accurate Clinical Management /ID# 159905, Baytown, Texas
  - Diagnostic Group Integrated He /ID# 159794, Beaumont, Texas
  - Arth and Osteo Clin Brazo Valley /ID# 163436, College Station, Texas
  - PCCR Solution /ID# 205723, Colleyville, Texas
  - Adriana Pop-Moody MD Clinic PA /ID# 159984, Corpus Christi, Texas
  - Metroplex Clinical Research /ID# 159785, Dallas, Texas
  - Rheumatic Disease Clin Res Ctr /ID# 161240, Houston, Texas
  - Rheumatology Clinic of Houston /ID# 161234, Houston, Texas
  - "DMCR-Texas Cent for Drug Dev /ID# 164191, Houston, Texas
  - West Texas Clinical Research /ID# 205722, Lubbock, Texas
  - P&I Clinical Research /ID# 159826, Lufkin, Texas
  - SW Rheumatology Res. LLC /ID# 159993, Mesquite, Texas
  - Trinity Universal Research Association /ID# 205721, Plano, Texas
  - Arthritis & Osteo Ctr of S. TX /ID# 163784, San Antonio, Texas
  - Arthritis Clinic of Central TX /ID# 164049, San Marcos, Texas
  - DM Clinical Research /ID# 161735, Tomball, Texas
  - Arthritis & Osteoporosis Clinic /ID# 159786, Waco, Texas
  - Arthritis Clinic of N. VA, P.C /ID# 159849, Arlington, Virginia
  - Ctr for Arth and Rheum Disease /ID# 159830, Chesapeake, Virginia
  - Swedish Medical Center /ID# 159890, Seattle, Washington
  - Arthritis Northwest, PLLC /ID# 166380, Spokane, Washington
  - West Virginia Research Inst /ID# 159791, South Charleston, West Virginia
  - Aurora Rheumatology and Immunotherapy Center /ID# 160043, Franklin, Wisconsin
- Argentina (9):
  - Centro Medico Privado/Reuma /ID# 159775, San Miguel de Tucumán, Ciuadad Autonoma de Buenos Aires
  - Centro Integral de Medicina Respiratoria (CIMER) /ID# 211237, San Miguel de Tucumán, Tucumán Province
  - Organizacion Medica de Investigacion (OMI) /ID# 160118, Buenos Aires
  - Hospital General de Agudos Ram /ID# 164378, Buenos Aires
  - Psoriahue Med Interdisciplinar /ID# 160506, Buenos Aires
  - Inst. de Rehab. Psicofisica /ID# 165154, CABA
  - Instituto CAICI /ID# 160119, Rosario, Santa FE
  - Centro Integral de Medicina Re /ID# 160258, SAN Miguel de Tucuman, Latam
  - Centro de Enfermedades del Hígado y Aparato Digestivo /ID# 165795, Santa Fe
- Australia (4):
  - Emeritus Research Sydney /ID# 166780, Botany, New South Wales
  - The Queen Elizabeth Hospital /ID# 169333, Woodville, South Australia
  - Barwon Rheumatology /ID# 166782, Geelong, Victoria
  - Heidelberg Repatriation Hospital /ID# 167450, Heidelberg West, Victoria
- Belarus (3):
  - Brest Regional Hospital /ID# 164535, Brest
  - Healthcare Institution /ID# 164536, Grodno
  - First City Clinical Hospital /ID# 164534, Minsk
- Reuma clinic /ID# 164243, Genk, Belgium
- Bosnia and Herzegovina (3):
  - University Clinical Centre of the Republic of Srpska /ID# 164503, Banja Luka, Republika Srpska
  - University Clinical Hospital Mostar /ID# 165799, Mostar
  - Clinical Center University of Sarajevo /ID# 164502, Sarajevo
- Brazil (11):
  - Instituto de Ciencias Farmacêuticas /ID# 163274, Aparecida de Goiânia, Goiás
  - CIP - Centro Internacional de Pesquisa /ID# 161821, Goiânia, Goiás
  - CMiP - Centro Mineiro de Pesquisa Ltda - ME /ID# 161819, Juiz de Fora, Minas Gerais
  - EDUMED Educacao em Saude S/S L /ID# 161816, Curitiba, Paraná
  - Instituto de Educação e Pesquisa do Hospital Moinhos de Vento /ID# 161813, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre /ID# 161820, Porto Alegre, Rio Grande do Sul
  - LMK Sevicos Medicos S/S /ID# 161812, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirão Preto - USP /ID# 163273, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC /ID# 163491, Santo André, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos do ABC /ID# 161810, Santo André, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas /ID# 161818, São Paulo
- Bulgaria (7):
  - Department of Rheumatology, Mu /ID# 169606, Plovdiv
  - Excelsior Medical Center /ID# 169609, Sofia
  - Multiprofile Hospital for Active Treatment - Sofia at Military Medical Academy /ID# 169608, Sofia
  - UMHAT Sv. Ivan Rilski /ID# 202393, Sofia
  - Medical Centre Synexus Sofia /ID# 202394, Sofia
  - Medical Centre Synexus Sofia, branch Stara Zagora /ID# 202524, Stara Zagora
  - Diagnostic Consultative Center /ID# 169607, Varna
- Canada (6):
  - Percuro Clinical Research, Ltd /ID# 157823, Victoria, British Columbia
  - Manitoba Clinic /ID# 157829, Winnipeg, Manitoba
  - Ciads /Id# 157831, Winnipeg, Manitoba
  - The Waterside Clinic /ID# 157826, Barrie, Ontario
  - Groupe de Recherche en Maladies Osseuses Inc /ID# 157824, Sainte-Foy, Quebec
  - Ctr. de Recherche Musculo-Sque /ID# 207069, Trois-Rivières, Quebec
- Chile (5):
  - M y F Estudios Clínicos Ltda. /ID# 168722, Ñuñoa, Santiago Metropolitan
  - CTR Estudios SpA /ID# 206217, Providencia
  - Centro Inter Estud Clin CIEC /ID# 168725, Santiago
  - Prosalud Ltda. /ID# 169546, Santiago
  - Clinica Dermacross S.A /ID# 168726, Vitacura Santiago
- China (15):
  - 1st Aff Hosp of Bengbu Medical College /ID# 201021, Bengbu, Anhui
  - Peking University Third Hospital /ID# 201973, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Shantou University Medical College /ID# 203371, Shantou, Guangdong
  - Zhuzhou Central Hospital /ID# 200201, Zhuzhou, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Monggolia Univers /ID# 171204, Baotou, Inner Mongolia
  - The First People's Hospital of Linyi /ID# 201970, Linyi, Shandong
  - Huashan Hospital of Fudan University /ID# 202191, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital /ID# 200202, Shanghai, Shanghai Municipality
  - West China Hospital /ID# 200199, Chengdu, Sichuan
  - Ningbo First Hospital /ID# 201874, Ningbo, Zhejiang
  - The Aff Hosp Inner Mongolia /ID# 207787, Hohhot
  - First Affiliated Hospital of Kunming Medical University /ID# 201264, Kunming
  - Affiliated hospital of nantong university /ID# 208234, Nantong
  - The First Affiliated Hospital of Soochow University /ID# 201875, Suzhou
  - People's Hospital of Xinjiang /ID# 201592, Ürümqi
- Colombia (5):
  - Centro de Investigacion en Reumatologia CIREEM /ID# 166030, Bogota, Cundinamarca
  - Fundacion Centro de Investigac /Id# 168201, Antioquia
  - Ctr Int de Reum del Caribe SAS /ID# 164051, Barranquilla
  - Preventive Care Sas /Id# 163781, Chía
  - Hospital Pablo Tobon Uribe /ID# 164233, Medellín
- Croatia (4):
  - Poliklinika Repromed /ID# 203555, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Rijeka /ID# 161159, Rijeka, Primorje-Gorski Kotar County
  - Medical Center Kuna-Peric /ID# 161160, Zagreb
  - Poliklinika Bonifarm /ID# 206662, Zagreb
- Czechia (5):
  - Revmatologicka ambulance /ID# 159637, Prague, Praha 4
  - Revmatologicka ambulance /ID# 159671, Prague, Praha 4
  - Revmatologie Bruntal, s.r.o /ID# 159636, Bruntál
  - Artroscan s.r.o. /ID# 159634, Ostrava
  - Medical Plus, s.r.o. /ID# 159635, Uherské Hradište
- Estonia (3):
  - Center of Clinical and Basic Research /ID# 163870, Tallinn, Harju
  - MediTrials /ID# 163706, Tartu, Tartu
  - East Tallinn Central Hospital /ID# 163790, Tallinn
- Germany (8):
  - Rheumazentrum Ruhrgebiet /ID# 163930, Herne, North Rhine-Westphalia
  - Immanuel-Krankenhaus /ID# 163931, Buch
  - University Clinic Carl Gustav /ID# 163926, Dresden
  - Polikilinik fuer Rheumatologie /ID# 163933, Düsseldorf
  - Cent fur Innovative Diagnostik /ID# 163927, Frankfurt
  - Hamburger Rheuma Forschungszentrum II im MVZ Rheumatologie und Autoimmunmedizin /ID# 204421, Hamburg
  - Dr. med. Jochen Walter FA fuer /ID# 168638, Rendsburg
  - Med. Universitaetsklinik Inner /ID# 163929, Tübingen
- Greece (6):
  - General Hospital of Athens Laiko /ID# 163476, Athens, Attica
  - General Hospital of Athens Laiko /ID# 163478, Athens, Attica
  - University General Hospital Attikon /ID# 163477, Athens, Attica
  - Naval Hospital of Athens /ID# 163486, Athens
  - University General Hospital of Heraklion PA.G.N.I /ID# 163472, Heraklion
  - Reg Gen Univ Hosp Larissa /ID# 163496, Larissa
- Hong Kong (3):
  - Prince of Wales Hospital /ID# 163506, Hong Kong
  - Queen Mary Hospital /ID# 162492, Hong Kong
  - Tuen Mun Hospital /ID# 162493, Tuenmen
- Hungary (10):
  - Synexus Magyarorszag Kft. - Gyula DRS /ID# 202209, Gyula, Bekes County
  - Qualiclinic Kft. /ID# 163278, Budapest III, Pest County
  - Szabolcs-Szatmar-Bereg Megyei Korhazak & Egyetemi Oktatok.- Klinikai Kutatasi O. /ID# 202584, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Synexus Magyarorszag Kft. - Zalaegerszeg AS /ID# 201884, Zalaegerszeg, Zala County
  - Betegapolo Irgalmas Rend - Budai Irgalmasrendi Korhaz /ID# 170719, Budapest
  - Revita Reumatologiai Rendelo /ID# 163277, Budapest
  - Obudai Egeszsegugyi Centrum Kft. /ID# 163279, Budapest
  - Synexus Magyarorszag Kft. /ID# 203012, Budapest
  - Debreceni Egyetem Kenezy Gyula /ID# 163276, Debrecen
  - Vital Medical Center Orvosi-es Fogaszati Kozpont /ID# 163275, Veszprém
- Ireland (2):
  - St Vincent's University Hosp /ID# 161073, Dublin
  - Croom Orthopaedic Hospital /ID# 164998, Limerick
- Israel (3):
  - Tel Aviv Sourasky Medical Center /ID# 169845, Tel Aviv, Tel Aviv
  - The Lady Davis Carmel MC /ID# 170262, Haifa
  - Sheba Medical Center /ID# 202532, Ramat Gan
- Italy (5):
  - AOU Federico II /ID# 202411, Naples, Campania
  - Azienda Unita Sanitaria Locale/IRCCS c/o Arcispedale Santa Maria Nuova /ID# 161090, Reggio Emilia, Emilia-Romagna
  - Policlinico Universitario Campus Bio-Medico /ID# 162306, Rome, Lazio
  - Ospedali Riuniti Universita /ID# 161085, Ancona
  - Azienda Ospedaliera Universitaria Policlinico "G. Rodolico - San Marco" /Id# 161084, Catania
- Japan (6):
  - Nagoya City University Hospital /ID# 162564, Nagoya, Aichi-ken
  - Fukuoka University Hospital /ID# 162086, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health /ID# 161473, Kitakyushu-shi, Fukuoka
  - Mie University Hospital /ID# 162080, Tsu, Mie-ken
  - National Hospital Organization Osaka Minami Medical Center /ID# 162590, Kawachinagano-shi, Osaka
  - St.Luke's International Hospital /ID# 162016, Chuo-ku, Tokyo
- Latvia (4):
  - M &M Centrs /Id# 161483, Ādaži
  - D.Saulites-Kandevicas PP in Cardiology and Rheumatology /ID# 161488, Liepāja
  - Clinic ORTO /ID# 161486, Riga
  - P. Stradins Clinical Univ Hosp /ID# 164442, Riga
- Lithuania (4):
  - VAKK dr. Kildos Clinic /ID# 167257, Kaunas
  - Klaipeda University Hospital /ID# 167258, Klaipėda
  - Public Institution Republican /ID# 165155, Šiauliai
  - Vilnius University Hospital /ID# 165123, Vilnius
- Malaysia (2):
  - Hospital Raja Permaisuri Bainun /ID# 161099, Ipoh, Perak
  - Hospital Tuanku Ja afar /ID# 161096, Seremban
- Mexico (3):
  - Instituto Jalisciense de Metabolismo SC /ID# 164005, Guadalajara, Jalisco
  - CINTRE, Centro de Investigación y Tratamiento Reumatológico SC /ID# 164006, Mexico City, Mexico City
  - Invest y Biomed de Chihuahua /ID# 164007, Chihuahua City
- Netherlands (3):
  - Medisch Centrum Leeuwarden /ID# 161575, Leeuwarden
  - Erasmus Medisch Centrum /ID# 161092, Rotterdam
  - Maasstad Ziekenhuis /ID# 160168, Rotterdam
- New Zealand (5):
  - Waikato Hospital /ID# 166415, Hamilton, Waikato Region
  - North Shore Hospital /ID# 169409, Auckland
  - Middlemore Hospital /ID# 166414, Auckland
  - Porter Rheumatology Ltd /ID# 200421, Nelson
  - Timaru Rheumatology Studies /ID# 166413, Timaru
- Norway (2):
  - Helse Forde /ID# 167853, Førde, Sogn Og Fjordane
  - St. Olavs Hospital HF /ID# 163321, Trondheim, Sor-Trondelag
- Poland (14):
  - NZOZ Nasz Lekarz /ID# 163774, Torun, Kuyavian-Pomeranian Voivodeship
  - Malopolskie Centrum Kliniczne /ID# 163777, Krakow, Lesser Poland Voivodeship
  - Synexus Polska Sp. z o.o. /ID# 204506, Wroclaw, Lower Silesian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku /ID# 206299, Gdansk, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni /ID# 207157, Gdynia, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial Katowice /ID# 204510, Katowice, Silesian Voivodeship
  - ETYKA-Osrodek Badan Klinicznyc /ID# 163776, Olsztyn, Warmian-Masurian Voivodeship
  - Centrum Kliniczno-Badawcze /ID# 161830, Elblag
  - Krakowskie Centrum Medyczne /ID# 206302, Krakow
  - Synexus Polska Sp. z o.o. Oddzial w Poznaniu /ID# 207158, Poznan
  - Medycyna Kliniczna /ID# 166288, Warsaw
  - Synexus Polska Sp. z.o.o. /ID# 203987, Warsaw
  - Reumatika - Centrum Reumatologii NZOZ /ID# 161831, Warsaw
  - Salve Medica Sp. z o.o. S.K. /ID# 206300, Lodz, Łódź Voivodeship
- Portugal (7):
  - Instituto Portugues De Reumatologia /ID# 165858, Lisbon, Lisbon District
  - Centro Hospitalar Lisboa Ocidental, EPE /ID# 165861, Lisbon, Lisbon District
  - Centro Hospitalar de Vila Nova Gaia/Espinho, EPE /ID# 165862, Vila Nova de Gaia, Porto District
  - Centro Hospitalar Lisboa Norte, EPE /ID# 165860, Lisbon
  - Hospital CUF Descobertas /ID# 165866, Lisbon
  - Hospital Beatriz Angelo /ID# 165865, Loures
  - Unidade Local De Saude Do Alto Minho /ID# 165863, Viana do Castelo
- Puerto Rico (3):
  - Cruz-Santana, Carolina, PR /ID# 163307, Carolina
  - Ponce Medical School Foundation /ID# 163920, Ponce
  - GCM Medical Group, PSC /ID# 162160, San Juan
- Russia (5):
  - Family Outpatient clinic#4 LLC /ID# 164530, Korolev, Moscow
  - LLC Medical Center /ID# 164529, Novosibirsk, Novosibirsk Oblast
  - Kazan State Medical University /ID# 164531, Kazan', Tatarstan, Respublika
  - Moscow S.P.Botkin City Clinica /ID# 164533, Moscow
  - State budgetary institution /ID# 164532, Saint Petersburg
- Serbia (5):
  - Institute for Rheumatology /ID# 166217, Belgrade, Beograd
  - Institute for Rheumatology /ID# 166223, Belgrade, Beograd
  - Institute for Rheumatology /ID# 166229, Belgrade, Beograd
  - Institute for Rheumatology /ID# 166231, Belgrade, Beograd
  - Military Medical Academy /ID# 166293, Belgrade, Beograd
- Singapore (2):
  - Singapore General Hospital /ID# 161094, Singapore, Central Singapore
  - Tan Tock Seng Hospital /ID# 161095, Singapore
- Slovakia (3):
  - MEDMAN s.r.o. /ID# 165892, Martin
  - Reumatologická ambulancia Reum.hapi s.r.o. /ID# 166486, Nové Mesto nad Váhom
  - Slovak research center Team Member, Thermium s.r.o. /ID# 166489, Pieštany
- Slovenia (3):
  - Univ Medical Ctr Ljubljana /ID# 164212, Ljubljana
  - University Medical Ctr Maribor /ID# 169260, Maribor
  - General Hospital Murska Sobota /ID# 164211, Murska Sobota
- South Africa (6):
  - Greenacres Hospital /ID# 164190, Port Elizabeth, Eastern Cape
  - Wits Clinical Research Site /ID# 163919, Johannesburg, Gauteng
  - University of Pretoria /ID# 163852, Pretoria, Gauteng
  - Jakaranda Hospital /ID# 164242, Pretoria, Gauteng
  - Arthritis Clinical Research Tr /ID# 163855, Cape Town, Western Cape
  - Winelands Medical Research Ctr /ID# 163853, Stellenbosch, Western Cape
- South Korea (2):
  - Ajou University Hospital /ID# 163891, Suwon, Gyeonggido
  - Inha University Hospital /ID# 163890, Junggu, Incheon Gwang Yeogsi
- Spain (4):
  - Hospital Universitario A Coruña - CHUAC /ID# 161129, A Coruña, A Coruna
  - Hospital Campus de la Salud /ID# 170760, Granada
  - Hospital Universitario Ramon y Cajal /ID# 161130, Madrid
  - Hospital Universitario 12 de Octubre /ID# 163198, Madrid
- Switzerland (2):
  - Kantonsspital St. Gallen /ID# 158131, Sankt Gallen, Canton of St. Gallen
  - HFR Fribourg - Hopital Canton /ID# 162090, Fribourg
- Taiwan (5):
  - China Medical University Hosp /ID# 159402, Taichung, Taichung
  - Chung Shan Medical University /ID# 159403, Taichung
  - National Taiwan University Hospital /ID# 160878, Taipei
  - Taipei Veterans General Hosp /ID# 166222, Taipei
  - Linkou Chang Gung Memorial Ho /ID# 166221, Taoyuan
- Turkey (Türkiye) (6):
  - Cukurova Universitesi Tip Fakultesi /ID# 162516, Saricam Adana, Adana
  - Hacettepe Universitesi Tip Fak /ID# 162518, Sihhiye, Ankara
  - Bakirkoy Dr. Sadi Konuk Training & Research Hospital /ID# 162517, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 163383, Istanbul
  - Necmettin Erbakan Universitesi /ID# 163382, Meram Konya
  - Sakarya Universitesi Egitim /ID# 163397, Sakarya
- Ukraine (11):
  - State Institution L. T. Malaya Therapy National Institution of NAMS of Ukraine /ID# 164170, Kharkiv, Kharkivs’ka Oblast’
  - Lviv Regional Clinical Hospita /ID# 164178, Lviv, Lviv Oblast
  - Kharkiv Regional Council Regional Clinical Hospital /ID# 210189, Kharkiv
  - NSC Strazhesko Ist Cardiology /ID# 164043, Kiev
  - Med Ctr of Private High Ed Ins /ID# 208527, Kyiv
  - Medical Center of LLC Medbud-Clinic /ID# 208528, Kyiv
  - Kyiv Railway Clinical Hosp No.2 /ID# 208951, Kyiv
  - LLC Revmocentr /ID# 164177, Kyiv
  - MNI KRC Kyiv Regional Clinical Hospital /ID# 210188, Kyiv
  - Odessa National Medical Univ /ID# 164244, Odesa
  - Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrogov /ID# 164245, Vinnytsia
- United Kingdom (6):
  - Whipps Cross Univ Hospital /ID# 161055, London, London, City of
  - Guy's and St Thomas' NHS Found /ID# 161065, London, London, City of
  - Christchurch Hospital /ID# 162702, Christchurch
  - UH Coventry & Warwickshire /ID# 162701, Coventry
  - Glasgow Royal Infirmary /ID# 162703, Glasgow
  - Luton & Dunstable University Hospital /ID# 162704, Luton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Burmester GR, Stigler J, Rubbert-Roth A, Tanaka Y, Azevedo VF, Coombs D, Lagunes I, Lippe R, Wung P, Gensler LS. Safety Profile of Upadacitinib up to 5 Years in Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis: An Integrated Analysis of Clinical Trials. Rheumatol Ther. 2024 Jun;11(3):737-753. doi: 10.1007/s40744-024-00671-4. Epub 2024 Apr 29. PMID 38683479
- [Derived] Cantini F, Marchesoni A, Novelli L, Gualberti G, Marando F, McDearmon-Blondell EL, Gao T, McGonagle D, Salvarani C. Effects of upadacitinib on enthesitis in patients with psoriatic arthritis: a post hoc analysis of SELECT-PsA 1 and 2 trials. Rheumatology (Oxford). 2024 Nov 1;63(11):3146-3154. doi: 10.1093/rheumatology/keae057. PMID 38331400
- [Derived] Rubbert-Roth A, Kakehasi AM, Takeuchi T, Schmalzing M, Palac H, Coombs D, Liu J, Anyanwu SI, Lippe R, Curtis JR. Malignancy in the Upadacitinib Clinical Trials for Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis. Rheumatol Ther. 2024 Feb;11(1):97-112. doi: 10.1007/s40744-023-00621-6. Epub 2023 Nov 20. PMID 37982966
- [Derived] Charles-Schoeman C, Choy E, McInnes IB, Mysler E, Nash P, Yamaoka K, Lippe R, Khan N, Shmagel AK, Palac H, Suboticki J, Curtis JR. MACE and VTE across upadacitinib clinical trial programmes in rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. RMD Open. 2023 Nov;9(4):e003392. doi: 10.1136/rmdopen-2023-003392. PMID 37945286
- [Derived] Baraliakos X, Ranza R, Ostor A, Ciccia F, Coates LC, Rednic S, Walsh JA, Douglas K, Gao T, Kato K, Song IH, Ganz F, Deodhar A. Efficacy and safety of upadacitinib in patients with active psoriatic arthritis and axial involvement: results from two phase 3 studies. Arthritis Res Ther. 2023 Apr 10;25(1):56. doi: 10.1186/s13075-023-03027-5. PMID 37038159
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] McInnes IB, Kato K, Magrey M, Merola JF, Kishimoto M, Haaland D, Chen L, Duan Y, Liu J, Lippe R, Wung P. Efficacy and Safety of Upadacitinib in Patients with Psoriatic Arthritis: 2-Year Results from the Phase 3 SELECT-PsA 1 Study. Rheumatol Ther. 2023 Feb;10(1):275-292. doi: 10.1007/s40744-022-00499-w. Epub 2022 Oct 15. PMID 36243812
- [Derived] Mease P, Kavanaugh A, Gladman D, FitzGerald O, Soriano ER, Nash P, Feng D, Lertratanakul A, Douglas K, Lippe R, Gossec L. Disease Control with Upadacitinib in Patients with Psoriatic Arthritis: A Post Hoc Analysis of the Randomized, Placebo-Controlled SELECT-PsA 1 and 2 Phase 3 Trials. Rheumatol Ther. 2022 Aug;9(4):1181-1191. doi: 10.1007/s40744-022-00449-6. Epub 2022 May 23. PMID 35606663
- [Derived] Burmester GR, Winthrop K, Blanco R, Nash P, Goupille P, Azevedo VF, Salvarani C, Rubbert-Roth A, Lesser E, Lippe R, Lertratanakul A, Mccaskill RM, Liu J, Ruderman EM. Safety Profile of Upadacitinib up to 3 Years in Psoriatic Arthritis: An Integrated Analysis of Two Pivotal Phase 3 Trials. Rheumatol Ther. 2022 Apr;9(2):521-539. doi: 10.1007/s40744-021-00410-z. Epub 2021 Dec 30. PMID 34970731
- [Derived] Nash P, Richette P, Gossec L, Marchesoni A, Ritchlin C, Kato K, McDearmon-Blondell EL, Lesser E, McCaskill R, Feng D, Anderson JK, Ruderman EM. Upadacitinib as monotherapy and in combination with non-biologic disease-modifying antirheumatic drugs for psoriatic arthritis. Rheumatology (Oxford). 2022 Aug 3;61(8):3257-3268. doi: 10.1093/rheumatology/keab905. PMID 34864911
- [Derived] Strand V, Mease PJ, Soriano ER, Kishimoto M, Salvarani C, Saffore CD, Zueger P, McDearmon-Blondell E, Kato K, Gladman DD. Improvement in Patient-Reported Outcomes in Patients with Psoriatic Arthritis Treated with Upadacitinib Versus Placebo or Adalimumab: Results from SELECT-PsA 1. Rheumatol Ther. 2021 Dec;8(4):1789-1808. doi: 10.1007/s40744-021-00379-9. Epub 2021 Oct 12. PMID 34636026
- [Derived] Muensterman E, Engelhardt B, Gopalakrishnan S, Anderson JK, Mohamed MF. Upadacitinib pharmacokinetics and exposure-response analyses of efficacy and safety in psoriatic arthritis patients - Analyses of phase III clinical trials. Clin Transl Sci. 2022 Jan;15(1):267-278. doi: 10.1111/cts.13146. Epub 2021 Oct 27. PMID 34464029
- [Derived] McInnes IB, Anderson JK, Magrey M, Merola JF, Liu Y, Kishimoto M, Jeka S, Pacheco-Tena C, Wang X, Chen L, Zueger P, Liu J, Pangan AL, Behrens F. Trial of Upadacitinib and Adalimumab for Psoriatic Arthritis. N Engl J Med. 2021 Apr 1;384(13):1227-1239. doi: 10.1056/NEJMoa2022516. PMID 33789011
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 282 sites in 44 countries and was initiated in April 2017. Adults with active psoriatic arthritis (PsA) and a history of inadequate response or intolerance to at least one non-biologic disease modifying anti-rheumatic drug (DMARD) were eligible for enrollment.
Pre-assignment Details: Participants were randomized in a 1:1:2:2:2 ratio to one of five treatment groups. Randomization was stratified by extent of psoriasis (≥ 3% body surface area [BSA] or < 3% BSA), current use of at least 1 non-biologic DMARD, presence of dactylitis, and presence of enthesitis, except for participants from China and Japan, where randomization was stratified by extent of psoriasis (≥ 3% BSA or < 3% BSA) only.
Groups:
- Placebo / Upadacitinib 15 mg: Participants randomized to receive matching placebo to upadacitinib orally once a day (QD) for 24 weeks followed by upadacitinib 15 mg once daily for 32 weeks (Weeks 24 to 56), as well as matching placebo to adalimumab administered by subcutaneous injection every other week (EOW) from Weeks 1 to 56.
- Placebo / Upadacitinib 30 mg: Participants randomized to receive matching placebo to upadacitinib orally QD for 24 weeks followed by upadacitinib 30 mg once daily for 32 weeks (Weeks 24 to 56), in addition to matching placebo to adalimumab administered by subcutaneous injection EOW from Weeks 1 to 56.
- Adalimumab 40 mg: Participants randomized to receive adalimumab 40 mg by subcutaneous injection EOW and matching placebo to upadacitinib orally QD for 56 weeks.
- Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg orally QD and matching placebo to adalimumab by subcutaneous injection EOW for 56 weeks.
- Upadacitinib 30 mg: Participants randomized to receive upadacitinib 30 mg orally QD and matching placebo to adalimumab by subcutaneous injection EOW for 56 weeks.
- Placebo / Upadacitinib 15 mg Period 2 (Weeks 56 to 260): Participants randomized to receive matching placebo to upadacitinib orally once a day (QD) for 24 weeks followed by upadacitinib 15 mg orally once a day (QD) for 32 weeks (Weeks 24 to 56), as well as matching placebo to adalimumab administered by subcutaneous injection every other week (EOW) from Weeks 1 to 56 in Period 1. During Period 2 (Weeks 56 to 260) participants continued to receive upadacitinib 15 mg orally once a day (QD).
- Placebo / Upadacitinib 30 mg Period 2 (Weeks 56 to 260): Participants randomized to receive matching placebo to upadacitinib orally once a day (QD) for 24 weeks followed by upadacitinib 30 mg orally once a day (QD) for 32 weeks (Weeks 24 to 56), as well as matching placebo to adalimumab administered by subcutaneous injection every other week (EOW) from Weeks 1 to 56 in Period 1. During Period 2 (Weeks 56 to 260) participants continued to receive upadacitinib 30 mg orally once a day (QD).
- Adalimumab 40 mg Period 2 (Weeks 56 to 260): Participants randomized to receive adalimumab 40 mg by subcutaneous injection every other week (EOW) and matching placebo to upadacitinib orally once a day (QD) for 56 weeks in Period 1 who continued to receive 40 mg adalimumab EOW in Period 2 (Weeks 56 to 260).
- Upadacitinib 15 mg Period 2 (Weeks 56 to 260): Participants randomized to receive upadacitinib 15 mg orally once a day (QD) and matching placebo to adalimumab by subcutaneous injection EOW for 56 weeks in Period 1 who continued to receive 15 mg upadacitinib QD in Period 2 (Weeks 56 to 260).
- Upadacitinib 30 mg Period 2 (Weeks 56 to 260): Participants randomized to receive upadacitinib 30 mg orally once a day (QD) and matching placebo to adalimumab by subcutaneous injection every other week (EOW) for 56 weeks in Period 1 who continued to receive 30 mg upadacitinib QD in Period 2 (Weeks 56 to 260).
Period: Period 1 (Week 1 - 56)
Arm/Group | Placebo / Upadacitinib 15 mg | Placebo / Upadacitinib 30 mg | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg | Placebo / Upadacitinib 15 mg Period 2 (Weeks 56 to 260) | Placebo / Upadacitinib 30 mg Period 2 (Weeks 56 to 260) | Adalimumab 40 mg Period 2 (Weeks 56 to 260) | Upadacitinib 15 mg Period 2 (Weeks 56 to 260) | Upadacitinib 30 mg Period 2 (Weeks 56 to 260)
Started | 211 | 212 | 429 | 430 | 423 | 0 | 0 | 0 | 0 | 0
Completed (Completed Week 56 (Period 1)) | 177 | 178 | 370 | 379 | 366 | 0 | 0 | 0 | 0 | 0
Not Completed | 34 | 34 | 59 | 51 | 57 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 7 | 11 | 9 | 21 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 20 | 29 | 24 | 24 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 1 | 4 | 8 | 7 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 6 | 3 | 8 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19 Logistical Restrictions | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other, not specified | 2 | 3 | 7 | 6 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Did not receive study drug | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 Week 56 - 260)
Arm/Group | Placebo / Upadacitinib 15 mg | Placebo / Upadacitinib 30 mg | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg | Placebo / Upadacitinib 15 mg Period 2 (Weeks 56 to 260) | Placebo / Upadacitinib 30 mg Period 2 (Weeks 56 to 260) | Adalimumab 40 mg Period 2 (Weeks 56 to 260) | Upadacitinib 15 mg Period 2 (Weeks 56 to 260) | Upadacitinib 30 mg Period 2 (Weeks 56 to 260)
Started | 0 | 0 | 0 | 0 | 0 | 177 | 178 | 366 | 378 | 365
Completed | 0 | 0 | 0 | 0 | 0 | 131 | 121 | 268 | 272 | 269
Not Completed | 0 | 0 | 0 | 0 | 0 | 46 | 57 | 98 | 106 | 96
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 14 | 17 | 14 | 28 | 28
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 11 | 21 | 45 | 44 | 32
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 7 | 6 | 12 | 12 | 7
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 9 | 6 | 7
Not completed — COVIID-19 infection | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3
Not completed — COVID-19 Logistical Restrictions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Other, not specified | 0 | 0 | 0 | 0 | 0 | 10 | 7 | 17 | 12 | 18
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo / Upadacitinib 15 mg | Placebo / Upadacitinib 30 mg | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg | Total
Number analyzed (Participants) | 211 | 212 | 429 | 430 | 423 | 1705
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (12.25) | 50.8 (12.18) | 51.4 (12.04) | 51.6 (12.18) | 49.9 (12.41) | 50.8 (12.22)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 185 | 182 | 362 | 368 | 371 | 1468
  65 - < 75 years | 24 | 28 | 61 | 52 | 46 | 211
  ≥ 75 years | 2 | 2 | 6 | 10 | 6 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 113 | 222 | 239 | 236 | 908
  Male | 113 | 99 | 207 | 191 | 187 | 797
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 37 | 65 | 60 | 53 | 244
  Not Hispanic or Latino | 182 | 175 | 364 | 370 | 370 | 1461
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 190 | 187 | 375 | 387 | 377 | 1516
  Black or African American | 2 | 1 | 2 | 1 | 3 | 9
  American Indian/Alaska Native | 1 | 1 | 2 | 0 | 2 | 6
  Native Hawaiian or other Pacific Islander | 0 | 1 | 2 | 0 | 1 | 4
  Asian | 16 | 21 | 41 | 37 | 34 | 149
  Multiple | 2 | 1 | 7 | 5 | 6 | 21
Extent of Psoriasis [Count of Participants; unit: Participants] — The extent of psoriasis was measured by the physician as the total body surface area (BSA) involved with psoriasis. For purposes of clinical estimation, the total surface of the participant's palm and five digits was assumed to be approximately equivalent to 1% of BSA.
  Participants
    < 3% BSA | 108 | 104 | 218 | 215 | 213 | 858
    ≥ 3% BSA | 103 | 108 | 211 | 214 | 210 | 846
    Missing | 0 | 0 | 0 | 1 | 0 | 1
Current Use of at Least 1 Non-Biologic DMARD [Count of Participants; unit: Participants]
  Yes | 174 | 173 | 346 | 353 | 345 | 1391
  No | 37 | 39 | 83 | 77 | 78 | 314
Presence of Dactylitis [Count of Participants; unit: Participants] — Dactylitis is characterized by swelling of the fingers or toes. The Leeds dactylitis index (LDI) is a score based on finger circumference and tenderness, assessed across all digits. The presence of a dactylitic digit is defined as at least 1 affected AND tender digit with circumference increase over reference digit ≥ 10%. Digit scores are calculated from the ratio of circumference between an affected digit and control digit and the tenderness score; unaffected digits have score = 0. Scores from each digit are summed to provide the final LDI.
  The presence of dactylitis is defined as LDI > 0.
  Participants
    Yes | 65 | 61 | 127 | 136 | 127 | 516
    No | 146 | 151 | 302 | 293 | 296 | 1188
    Missing | 0 | 0 | 0 | 1 | 0 | 1
Presence of Enthesitis [Count of Participants; unit: Participants] — Enthesitis is inflammation of the entheses, the specific point where tendons or ligaments attach to bone. Tenderness at 9 bilateral sites was assessed as present (1) or absent (0). The total enthesitis count is calculated by summing the tenderness scores from all 18 sites (range 0 - 18).
  Presence of enthesitis is defined as Total Enthesitis Count > 0.
  Participants
    Yes | 161 | 161 | 331 | 333 | 331 | 1317
    No | 50 | 51 | 98 | 96 | 92 | 387
    Missing | 0 | 0 | 0 | 1 | 0 | 1
Duration of Psoriatic Arthritis Symptoms [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 211 | 212 | 428 | 429 | 423 | 1703
    (all) | 9.6 (9.00) | 9.0 (8.15) | 9.1 (8.78) | 9.2 (8.63) | 9.2 (8.28) | 9.2 (8.56)
Duration of PsA Diagnosis [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 211 | 212 | 429 | 429 | 423 | 1704
    (all) | 6.4 (7.39) | 6.1 (6.63) | 5.9 (7.06) | 6.2 (7.41) | 5.9 (6.37) | 6.1 (6.97)
Tender Joint Count (TJC) [Mean (Standard Deviation); unit: joints] — A total of 68 joints were assessed for the presence or absence of tenderness. Population: Participants with available data
  joints
    number analyzed (Participants) | 211 | 212 | 429 | 429 | 423 | 1704
    (all) | 20.7 (15.67) | 19.3 (12.89) | 20.1 (13.82) | 20.4 (14.72) | 19.4 (13.32) | 20.0 (14.06)
Swollen Joint Count (SJC) [Mean (Standard Deviation); unit: joints] — A total of 66 joints were assessed for the presence or absence of swelling. Population: Participants with available data
  joints
    number analyzed (Participants) | 211 | 212 | 429 | 429 | 423 | 1704
    (all) | 11.4 (8.47) | 10.7 (7.85) | 11.6 (8.75) | 11.6 (9.31) | 10.6 (7.06) | 11.2 (8.37)
Patient's Assessment of Pain [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to indicate the severity of their arthritis pain within the previous week on a numeric rating scale (NRS) from 0 to 10. A score of 0 indicates "no pain" and a score of 10 indicates "worst possible pain." Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 211 | 210 | 428 | 425 | 421 | 1695
    (all) | 6.0 (2.21) | 6.2 (2.07) | 6.0 (2.08) | 6.2 (2.07) | 5.9 (2.05) | 6.0 (2.09)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: units on a scale] — The participant was asked to rate their current psoriatic arthritis disease activity on a 0 to 10 NRS, where 0 indicates very low disease activity and 10 indicates very high disease activity. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 211 | 210 | 428 | 425 | 421 | 1695
    (all) | 6.2 (2.17) | 6.4 (1.89) | 6.3 (2.03) | 6.6 (2.03) | 6.4 (2.07) | 6.4 (2.04)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: units on a scale] — The physician rated the participant's current global psoriatic arthritis disease activity (independently from the participant's assessment) on a 0 to 10 NRS where 0 indicates very low disease activity and 10 indicates very high disease activity. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 211 | 212 | 429 | 429 | 423 | 1704
    (all) | 6.6 (1.65) | 6.4 (1.62) | 6.6 (1.65) | 6.7 (1.62) | 6.5 (1.68) | 6.5 (1.65)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 211 | 210 | 428 | 425 | 421 | 1695
    (all) | 1.08 (0.638) | 1.15 (0.640) | 1.12 (0.626) | 1.15 (0.653) | 1.09 (0.630) | 1.12 (0.637)
High-sensitivity C-reactive Protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] — C-reactive protein (CRP) is a protein found in blood. CRP levels rise in response to inflammation. Population: Participants with available data
  mg/L
    number analyzed (Participants) | 211 | 212 | 429 | 429 | 423 | 1704
    (all) | 12.00 (17.146) | 10.96 (14.357) | 10.91 (15.462) | 11.00 (14.910) | 11.49 (15.355) | 11.22 (15.372)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom ACR data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants received matching placebo to upadacitinib orally QD and matching placebo to adalimumab SC EOW.
- Adalimumab 40 mg: Participants received adalimumab 40 mg SC EOW and matching placebo to upadacitinib orally QD.
- Upadacitinib 15 mg: Participants received upadacitinib 15 mg orally QD and matching placebo to adalimumab SC EOW.
- Upadacitinib 30 mg: Participants received upadacitinib 30 mg orally QD and matching placebo to adalimumab SC EOW.
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 423 | 429 | 429 | 423
percentage of participants | 36.2 [31.6 to 40.7] | 65.0 [60.5 to 69.5] | 70.6 [66.3 to 74.9] | 78.5 [74.6 to 82.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — The overall type I error rate of the primary and the 14 ranked secondary endpoints was controlled using a two-part sequential graphical multiple testing procedure starting with the primary endpoint using α/2 for each dose followed by a prespecified α transfer path; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 34.5, 95% CI 2-sided [28.2 to 40.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 42.3, 95% CI 2-sided [36.3 to 48.3] — Response Rate Difference = Upadacitinib - Placebo

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data; a mixed effect model repeat measurement (MMRM) analysis with longitudinal data from observed cases up to Week 12 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 392 | 406 | 404 | 398
units on a scale | -0.14 [-0.18 to -0.09] | -0.34 [-0.38 to -0.29] | -0.42 [-0.47 to -0.37] | -0.47 [-0.52 to -0.42]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; MMRM analysis including treatment, visit, treatment-by-visit interaction, current DMARD use (yes/no) as fixed factors and Baseline value as covariate; Least Squares (LS) Mean Difference = -0.28, 95% CI 2-sided [-0.35 to -0.22] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.34, 95% CI 2-sided [-0.40 to -0.27] — Treatment Difference = Upadacitinib - Placebo

3. Secondary Outcome: Percentage of Participants Achieving a Static Investigator Global Assessment (sIGA) of Psoriasis of 0 or 1 and at Least a 2-point Improvement From Baseline (sIGA 0/1) at Week 16
Description: The sIGA is a 5 point scale ranging from 0 to 4, based on the investigator's assessment of the average elevation, erythema, and scaling of all psoriatic lesions at the current visit. A lower score indicates less severe psoriasis (0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe).
Time Frame: Baseline and Week 16
Population: Full analysis set participants with a Baseline sIGA score ≥ 2; participants who prematurely discontinued from study drug prior to Week 16 or for whom sIGA data were missing at Week 16 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 313 | 330 | 322 | 324
percentage of participants | 10.9 [7.4 to 14.3] | 38.5 [33.2 to 43.7] | 41.9 [36.5 to 47.3] | 54.0 [48.6 to 59.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusting for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 31.1, 95% CI 2-sided [24.7 to 37.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusting for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 43.1, 95% CI 2-sided [36.7 to 49.6] — Response Rate Difference = Upadacitinib - Placebo

4. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 75 Response at Week 16
Description: PASI is a composite score based on the percentage of the body surface area (BSA) affected by psoriasis and the intensity of erythema (reddening), induration (thickening or hardening of the skin), and desquamation (peeling of the skin) of lesions assessed at 4 anatomic sites (head, upper extremities, trunk, and lower extremities). At each location, the percentage of BSA involvement is assigned a score from 0 (no involvement) to 6 (90% to 100% involvement), and erythema, induration, and desquamation are scored on a scale from 0 (no symptoms) to 4 (very marked).
  The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). A PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from Baseline in PASI score, and was assessed in participants with Baseline psoriasis BSA involvement ≥ 3%.
Time Frame: Baseline and Week 16
Population: Full analysis set participants with Baseline psoriasis BSA involvement ≥ 3%; participants who prematurely discontinued from study drug prior to Week 16 or for whom PASI data were missing at Week 16 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 211 | 211 | 214 | 210
percentage of participants | 21.3 [15.8 to 26.9] | 53.1 [46.3 to 59.8] | 62.6 [56.1 to 69.1] | 62.4 [55.8 to 68.9]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusting for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 41.3, 95% CI 2-sided [32.8 to 49.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 41.1, 95% CI 2-sided [32.5 to 49.6] — Response Rate Difference = Upadacitinib - Placebo

5. Secondary Outcome: Change From Baseline in Modified PsA Total Sharp/Van Der Heijde Score (mTSS) at Week 24
Description: The Sharp-van der Heijde modified scoring method for PsA measures the level of joint damage from radiographs of the hands and feet, and was assessed by 2 independent, blinded readers.
  Joint erosion severity was assessed in 20 joints in each hand and wrist and 6 joints in each foot. Each joint was scored from 0 (no erosion) to 5 for hands/wrists or to 10 for feet (complete collapse). The total erosion score ranges from 0 to 320 (worst).
  Joint space narrowing (JSN) was assessed in 20 joints of each hand and wrist, and 6 joints of each foot, from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation). The total JSN score ranges from 0 to 208 (worst).
  Joints with gross osteolysis or pencil in cup were assigned the maximum score for both erosions and JSN.
  The total mTSS score is the sum of the joint erosion and JSN scores and ranges from 0 (normal) to 528 (worst). A negative change from Baseline indicates improvement in joint damage.
Time Frame: Baseline and Week 24
Population: Full analysis set participants with available data at Baseline; linear extrapolation was used for participants who discontinued prior to Week 24 or who were rescued prior to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 372 | 384 | 391 | 383
score on a scale | 0.25 [0.13 to 0.36] | 0.01 [-0.11 to 0.13] | -0.04 [-0.16 to 0.07] | 0.03 [-0.08 to 0.15]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0002, ANCOVA; ANCOVA model including treatment and the stratification factor current DMARD use (yes/no) as fixed factors and Baseline value as covariate; LS Mean Difference = -0.29, 95% CI 2-sided [-0.44 to -0.14] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0069, ANCOVA; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = -0.21, 95% CI 2-sided [-0.36 to -0.06] — Treatment Difference = Upadacitinib - Placebo

6. Secondary Outcome: Percentage of Participants Achieving Minimal Disease Activity (MDA) at Week 24
Description: A participant was classified as achieving MDA if 5 of the following 7 criteria were met:
  * Tender joint count (out of 68 joints) ≤ 1
  * Swollen joint count (out of 66 joints) ≤ 1
  * PASI score ≤ 1 (score ranges from 0 - 72) or percent BSA involved with psoriasis ≤ 3%
  * Patient's assessment of pain ≤ 1.5 (NRS from 0 to 10)
  * Patient's Global Assessment of disease activity ≤ 2 (NRS from 0 to 10)
  * HAQ-DI score ≤ 0.5 (index score ranges from 0 to 3)
  * Leeds Enthesitis Index ≤ 1 (assesses the presence or absence of enthesitis at 3 bilateral sites, with an overall score range from 0 to 6)
Time Frame: Week 24
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 24 or for whom data were missing at Week 24, or who met the rescue criteria at Week 16 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 423 | 429 | 429 | 423
percentage of participants | 12.3 [9.2 to 15.4] | 33.3 [28.9 to 37.8] | 36.6 [32.0 to 41.2] | 45.4 [40.6 to 50.1]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 24.3, 95% CI 2-sided [18.8 to 29.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 33.1, 95% CI 2-sided [27.4 to 38.8] — Response Rate Difference = Upadacitinib - Placebo

7. Secondary Outcome: Percentage of Participants With Resolution of Enthesitis at Week 24
Description: Resolution of enthesitis is defined as a Leeds Enthesitis Index (LEI) score = 0.
  LEI is an enthesitis measure developed specifically for PsA and assesses the presence or absence of tenderness at the following 3 bilateral enthesial sites: medial femoral condyles, lateral epicondyles of the humerus, and Achilles tendon insertions. Tenderness on examination is recorded as either present (coded as 1), absent (coded as 0), or not assessed for each of the 6 sites. The LEI is calculated by taking the sum of the scores from the 6 sites. The LEI ranges from 0 to 6 (worst).
Time Frame: Week 24
Population: Full analysis set participants with a Baseline LEI > 0; participants who prematurely discontinued from study drug prior to Week 24 or for whom data were missing at Week 24, or who met the rescue criteria at Week 16 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 241 | 265 | 270 | 267
percentage of participants | 32.4 [26.5 to 38.3] | 47.2 [41.2 to 53.2] | 53.7 [47.8 to 59.7] | 57.7 [51.8 to 63.6]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 21.3, 95% CI 2-sided [13.0 to 29.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 25.3, 95% CI 2-sided [16.9 to 33.7] — Response Rate Difference = Upadacitinib - Placebo

8. Secondary Outcome: Percentage of Participants With an ACR20 Response at Week 12 - Non-inferiority Versus Adalimumab
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Adalimumab 40 mg: Participants received adalimumab 40 mg SC EOW and placebo to upadacitinib orally QD.
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 423 | 429 | 429 | 423
percentage of participants | 36.2 [31.6 to 40.7] | 65.0 [60.5 to 69.5] | 70.6 [66.3 to 74.9] | 78.5 [74.6 to 82.4]
Statistical Analysis 1: Comparison: Adalimumab 40 mg vs Upadacitinib 15 mg; Test type: Non-Inferiority — Non-inferiority of each upadacitinib dose versus adalimumab was assessed using Koch's 3-arm approach; non-inferiority was achieved if upadacitinib preserved at least 50% of the placebo-subtracted adalimumab effect. The overall type I error rate of the primary and the 14 ranked secondary endpoints was controlled using a two-part sequential graphical multiple testing procedure starting with the primary endpoint using α/2 for each dose followed by a prespecified α transfer path; p < 0.0001, Koch 3-Arm Test; Percent Adalimumab Effect Preservation = 119.381, 95% CI 2-sided [97.987 to 147.942] — The percent of adalimumab effect preservation is the point estimate of 3-arm non-inferiority analysis, which is calculated by (Upadacitinib - Placebo) / (Adalimumab - Placebo) * 100
Statistical Analysis 2: Comparison: Adalimumab 40 mg vs Upadacitinib 30 mg; Test type: Non-Inferiority — [test comment as in outcome 8, analysis 1]; p < 0.0001, Koch 3-Arm Test; Percent Adalimumab Effect Preservation = 146.604, 95% CI 2-sided [122.817 to 180.398] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Score (PCS) at Week 12
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component score is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 394 | 410 | 405 | 398
score on a scale | 3.19 [2.41 to 3.96] | 6.82 [6.07 to 7.58] | 7.86 [7.09 to 8.63] | 8.90 [8.13 to 9.68]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 4.67, 95% CI 2-sided [3.67 to 5.67] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 5.72, 95% CI 2-sided [4.71 to 6.72] — Treatment Difference = Upadacitinib - Placebo

10. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 12
Description: The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days, including physical fatigue (e.g., I feel tired), functional fatigue (e.g., trouble finishing things), emotional fatigue (e.g., frustration), and social consequences of fatigue (e.g., limits social activity). Participants respond to the questions on a scale from 0 'not at all' to 4 'very much'. The FACIT Fatigue score is computed by summing the item scores, after reversing those items that are worded in the negative direction. The FACIT-Fatigue subscale score ranges from 0 to 52, where higher scores represent less fatigue. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 394 | 410 | 404 | 398
score on a scale | 2.8 [1.9 to 3.7] | 5.7 [4.8 to 6.6] | 6.3 [5.4 to 7.2] | 7.1 [6.2 to 8.0]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 3.5, 95% CI 2-sided [2.4 to 4.7] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 4.3, 95% CI 2-sided [3.1 to 5.5] — Treatment Difference = Upadacitinib - Placebo

11. Secondary Outcome: Percentage of Participants With an ACR20 Response at Week 12 - Superiority Versus Adalimumab
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 423 | 429 | 429 | 423
percentage of participants | 36.2 [31.6 to 40.7] | 65.0 [60.5 to 69.5] | 70.6 [66.3 to 74.9] | 78.5 [74.6 to 82.4]
Statistical Analysis 1: Comparison: Adalimumab 40 mg vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0815, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusting for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 5.6, 95% CI 2-sided [-0.6 to 11.8] — Response Rate Difference = Upadacitinib - Adalimumab
Statistical Analysis 2: Comparison: Adalimumab 40 mg vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); LS Mean Difference = 13.5, 95% CI 2-sided [7.5 to 19.4] — Response Rate Difference = Upadacitinib - Adalimumab

12. Secondary Outcome: Percentage of Participants With Resolution of Dactylitis at Week 24
Description: Resolution of dactylitis is defined as a Leeds Dactylitis Index (LDI) score = 0.
  The Leeds Dactylitis Index (LDI) is a score based on finger circumference and tenderness, assessed and summed across all dactylitic digits (fingers and toes). The presence of a dactylitic digit is defined as at least one affected AND tender digit with circumference increase over reference digit ≥ 10%. The reference digit circumference is either the contralateral digit (unaffected digit on opposite hand or foot) if available, or from a standard reference table if otherwise. Tenderness of affected digits is assessed on a scale from 0 [none] to 3 [worst].
  The ratio of circumference between an affected digit and reference digit is multiplied by the tenderness score for each affected digit. The results from each involved digit are summed to provide the final LDI. A higher LDI indicates worse dactylitis.
Time Frame: Week 24
Population: Full analysis set participants with a Baseline LDI > 0; participants who prematurely discontinued from study drug prior to Week 24 or for whom data were missing at Week 24, or who met the rescue criteria at Week 16 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 126 | 127 | 136 | 127
percentage of participants | 39.7 [31.1 to 48.2] | 74.0 [66.4 to 81.6] | 76.5 [69.3 to 83.6] | 79.5 [72.5 to 86.5]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel — This comparison was not tested for statistical significance because the hierarchical testing procedures stopped at ACR 20 at Week 12 superiority test of upadacitinib 15 mg versus adalimumab 40 mg; Cochran-Mantel-Haenszel test adjusting for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 36.8, 95% CI 2-sided [25.7 to 47.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 39.8, 95% CI 2-sided [28.8 to 50.9] — Response Rate Difference = Upadacitinib - Placebo

13. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain - Superiority Versus Adalimumab
Description: Participants were asked to indicate the severity of their arthritis pain within the previous week on a numerical rating scale (NRS) from 0 to 10. A score of 0 indicates "no pain" and a score of 10 indicates "worst possible pain." A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 392 | 406 | 404 | 398
units on a scale | -0.9 [-1.2 to -0.7] | -2.3 [-2.5 to -2.1] | -2.3 [-2.5 to -2.0] | -2.7 [-2.9 to -2.5]
Statistical Analysis 1: Comparison: Adalimumab 40 mg vs Upadacitinib 15 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.8970, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.3] — Treatment Difference = Upadacitinib - Adalimumab
Statistical Analysis 2: Comparison: Adalimumab 40 mg vs Upadacitinib 30 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0028, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.2] — Treatment Difference = Upadacitinib - Adalimumab

14. Secondary Outcome: Change From Baseline in HAQ-DI - Superiority Versus Adalimumab
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 392 | 406 | 404 | 398
score on a scale | -0.14 [-0.18 to -0.09] | -0.34 [-0.38 to -0.29] | -0.42 [-0.47 to -0.37] | -0.47 [-0.52 to -0.42]
Statistical Analysis 1: Comparison: Adalimumab 40 mg vs Upadacitinib 15 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0162, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.08, 95% CI 2-sided [-0.15 to -0.01] — Treatment Difference = Upadacitinib - Adalimumab
Statistical Analysis 2: Comparison: Adalimumab 40 mg vs Upadacitinib 30 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.14, 95% CI 2-sided [-0.20 to -0.07] — Treatment Difference = Upadacitinib - Adalimumab

15. Secondary Outcome: Change From Baseline in Self-Assessment of Psoriasis Symptoms (SAPS) Questionnaire at Week 16
Description: The SAPS is an 11-item self-assessment of psoriasis symptoms that includes questions on: pain, itching, redness, scaling, flaking, bleeding, burning, stinging, tenderness, pain due to skin cracking, and joint pain. Each item is scored from 0 to 10, with 0 being least severe and 10 being most severe. The total score is generated by summing the 11 items and ranges from 0 to 110 (worst). A negative change from Baseline in the total score indicates improvement.
Time Frame: Baseline and Week 16
Population: Full analysis set participants with available data; a mixed effect model repeat measurement (MMRM) analysis with longitudinal data from observed cases up to Week 16 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 388 | 407 | 396 | 395
score on a scale | -8.2 [-10.2 to -6.3] | -22.7 [-24.7 to -20.8] | -25.3 [-27.3 to -23.4] | -28.1 [-30.0 to -26.1]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -17.1, 95% CI 2-sided [-19.6 to -14.6] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -19.8, 95% CI 2-sided [-22.3 to -17.3] — Treatment Difference = Upadacitinib - Placebo

16. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 423 | 429 | 429 | 423
percentage of participants | 13.2 [10.0 to 16.5] | 37.5 [32.9 to 42.1] | 37.5 [32.9 to 42.1] | 51.8 [47.0 to 56.5]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 24.3, 95% CI 2-sided [18.7 to 29.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusting for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 38.5, 95% CI 2-sided [32.8 to 44.3] — Response Rate Difference = Upadacitinib - Placebo

17. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 423 | 429 | 429 | 423
percentage of participants | 2.4 [0.9 to 3.8] | 13.8 [10.5 to 17.0] | 15.6 [12.2 to 19.1] | 25.3 [21.2 to 29.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusting for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 13.3, 95% CI 2-sided [9.5 to 17.0] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusting for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 22.9, 95% CI 2-sided [18.5 to 27.3] — Response Rate Difference = Upadacitinib - Placebo

18. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 2
Description: as for outcome 1
Time Frame: Baseline and Week 2
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 2 or for whom ACR data were missing at Week 2 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab 40 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 423 | 429 | 429 | 423
percentage of participants | 12.1 [9.0 to 15.2] | 30.3 [26.0 to 34.7] | 28.2 [23.9 to 32.5] | 38.3 [33.7 to 42.9]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusting for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 16.1, 95% CI 2-sided [10.9 to 21.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusting for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 26.2, 95% CI 2-sided [20.7 to 31.8] — Response Rate Difference = Upadacitinib - Placebo

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from time informed consent was signed to end of the study. Median time on follow-up in Period 1 (days): Upa 15 mg (415); Upa 30 mg (414); Ada 40 mg (194); Pbo up to Wk 24 (418); Pbo/Upa 15 mg Wk 24-56 (419); and Pbo/Upa 30 mg Wk 24-56 (776.5). Median time on follow-up in Period 2 (days): Upa 15 mg (1458); Upa 30 mg (796.5); Ada 40 mg (1486); Pbo/Upa 15 mg (1459); Pbo/Upa 30 mg (790.5); and Upa 30 mg/Upa 15 mg (842).
Groups:
- Upadacitinib 15 mg Period 1 (Weeks 1 to 56): Participants randomized to receive upadacitinib 15 mg orally once a day (QD) and matching placebo to adalimumab by subcutaneous injection every other week (EOW) for 56 weeks in Period 1.
- Upadacitinib 30 mg Period 1 (Weeks 1 to 56): Participants randomized to receive upadacitinib 30 mg orally once a day (QD) and matching placebo to adalimumab by subcutaneous injection every other week (EOW) for 56 weeks in Period 1.
- Adalimumab 40 mg Period 1 (Weeks 1 to 56): Participants randomized to receive adalimumab 40 mg by subcutaneous injection every other week (EOW) and matching placebo to upadacitinib orally once a day (QD) for 56 weeks in Period 1.
- Placebo Period 1 (Weeks 1 to 24): Participants randomized to receive matching placebo to upadacitinib orally once a day (QD) for 24 weeks, as well as matching placebo to adalimumab administered by subcutaneous injection every other week (EOW) from Weeks 1 to 24 in Period 1.
- Placebo / Upadacitinib 15 mg Period 1 (Weeks 24 to 56): Participants randomized to receive matching placebo to upadacitinib orally once a day (QD) for 24 weeks followed by upadacitinib 15 mg orally once a day (QD) for 32 weeks (Weeks 24 to 56), as well as matching placebo to adalimumab administered by subcutaneous injection every other week (EOW) from Weeks 1 to 56 in Period 1.
- Placebo / Upadacitinib 30 mg Period 1 (Weeks 24 to 56): Participants randomized to receive matching placebo to upadacitinib orally once a day (QD) for 24 weeks followed by upadacitinib 30 mg orally once a day (QD) for 32 weeks (Weeks 24 to 56), as well as matching placebo to adalimumab administered by subcutaneous injection every other week (EOW) from Weeks 1 to 56 in Period 1.
- Upadacitinib 30 mg / Upadacitinib 15 mg Period 2 (Weeks 56 to 260): Participants randomized to receive upadacitinib 30 mg orally once a day (QD) who were switched to upadacitinib 15 mg orally once a day (QD) at their next scheduled study visit in Period 2 after Protocol Amendment 7 was approved (30 January 2021).
Arm/Group | Upadacitinib 15 mg Period 1 (Weeks 1 to 56) | Upadacitinib 30 mg Period 1 (Weeks 1 to 56) | Adalimumab 40 mg Period 1 (Weeks 1 to 56) | Placebo Period 1 (Weeks 1 to 24) | Placebo / Upadacitinib 15 mg Period 1 (Weeks 24 to 56) | Placebo / Upadacitinib 30 mg Period 1 (Weeks 24 to 56) | Upadacitinib 15 mg Period 2 (Weeks 56 to 260) | Upadacitinib 30 mg Period 2 (Weeks 56 to 260) | Adalimumab 40 mg Period 2 (Weeks 56 to 260) | Placebo / Upadacitinib 15 mg Period 2 (Weeks 56 to 260) | Placebo / Upadacitinib 30 mg Period 2 (Weeks 56 to 260) | Upadacitinib 30 mg / Upadacitinib 15 mg Period 2 (Weeks 56 to 260)
All-Cause Mortality (participants affected / at risk) | 3/430 | 1/423 | 1/429 | 1/423 | 0/188 | 0/190 | 14/378 | 8/366 | 4/366 | 3/177 | 3/178 | 6/443
Serious Adverse Events (participants affected / at risk) | 28/430 | 46/423 | 35/429 | 13/423 | 10/188 | 11/190 | 109/378 | 66/366 | 73/366 | 34/177 | 25/178 | 55/443
Other Adverse Events (participants affected / at risk) | 247/430 | 262/423 | 220/429 | 150/423 | 61/188 | 76/190 | 277/378 | 218/366 | 246/366 | 130/177 | 114/178 | 271/443
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Upadacitinib 15 mg Period 1 (Weeks 1 to 56) (N=430) | Upadacitinib 30 mg Period 1 (Weeks 1 to 56) (N=423) | Adalimumab 40 mg Period 1 (Weeks 1 to 56) (N=429) | Placebo Period 1 (Weeks 1 to 24) (N=423) | Placebo / Upadacitinib 15 mg Period 1 (Weeks 24 to 56) (N=188) | Placebo / Upadacitinib 30 mg Period 1 (Weeks 24 to 56) (N=190) | Upadacitinib 15 mg Period 2 (Weeks 56 to 260) (N=378) | Upadacitinib 30 mg Period 2 (Weeks 56 to 260) (N=366) | Adalimumab 40 mg Period 2 (Weeks 56 to 260) (N=366) | Placebo / Upadacitinib 15 mg Period 2 (Weeks 56 to 260) (N=177) | Placebo / Upadacitinib 30 mg Period 2 (Weeks 56 to 260) (N=178) | Upadacitinib 30 mg / Upadacitinib 15 mg Period 2 (Weeks 56 to 260) (N=443)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAEMIA MACROCYTIC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOID TISSUE HYPERPLASIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AORTIC VALVE STENOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC DISORDER (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHRONIC CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAROXYSMAL ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HYDROCELE (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GOITRE (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIPLOPIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYELID PTOSIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL STRANGULATED HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FAECALOMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRIC ULCER PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRODUODENAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIATUS HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGEAL SPASM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CYST RUPTURE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DROWNING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RETENTION CYST (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IMMUNE SYSTEM DISORDER (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BONE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (12) | 8 (9) | 4 (4) | 1 (1) | 1 (1) | 4 (4)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 18 (20) | 16 (20) | 3 (4) | 8 (9) | 6 (8) | 5 (7)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CHRONIC TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS INTESTINAL PERFORATED (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
H1N1 INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTED DERMAL CYST (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 7 (7) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
PNEUMONIA ACINETOBACTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SALPINGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPUTUM PURULENT (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TUBERCULOUS PLEURISY (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CHEST INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL FOREIGN BODY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OPTIC NERVE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SOFT TISSUE FOREIGN BODY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STRESS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRAUMATIC LIVER INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CORTISOL ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FRUCTOSE INTOLERANCE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FACET JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
FRACTURE NONUNION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JAW DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (4) | 5 (6) | 1 (2) | 1 (2) | 5 (5)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SNAPPING HIP SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL RETROLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CLEAR CELL RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMANGIOMA OF LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HORMONE RECEPTOR POSITIVE HER2 NEGATIVE BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INVASIVE BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
LARYNGEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYELOFIBROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUROENDOCRINE CARCINOMA OF THE SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POORLY DIFFERENTIATED THYROID CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCHWANNOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THYROID ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CERVICAL RADICULOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEMYELINATION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETIC NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LACUNAR STROKE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NERVE COMPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
VITH NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UNINTENDED PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BIPOLAR I DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BIPOLAR DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CALCULUS URINARY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URETHRAL STENOSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CERVICAL POLYP (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL HYPERTROPHY (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALLOPIAN TUBE CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FIBROCYSTIC BREAST DISEASE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHAGIC OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OVARIAN STROMAL HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE POLYP (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ASPHYXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OBSTRUCTIVE SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONSILLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS EXFOLIATIVE GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATOMYOSITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUPERFICIAL VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VARICOSE VEIN (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Upadacitinib 15 mg Period 1 (Weeks 1 to 56) (N=430) | Upadacitinib 30 mg Period 1 (Weeks 1 to 56) (N=423) | Adalimumab 40 mg Period 1 (Weeks 1 to 56) (N=429) | Placebo Period 1 (Weeks 1 to 24) (N=423) | Placebo / Upadacitinib 15 mg Period 1 (Weeks 24 to 56) (N=188) | Placebo / Upadacitinib 30 mg Period 1 (Weeks 24 to 56) (N=190) | Upadacitinib 15 mg Period 2 (Weeks 56 to 260) (N=378) | Upadacitinib 30 mg Period 2 (Weeks 56 to 260) (N=366) | Adalimumab 40 mg Period 2 (Weeks 56 to 260) (N=366) | Placebo / Upadacitinib 15 mg Period 2 (Weeks 56 to 260) (N=177) | Placebo / Upadacitinib 30 mg Period 2 (Weeks 56 to 260) (N=178) | Upadacitinib 30 mg / Upadacitinib 15 mg Period 2 (Weeks 56 to 260) (N=443)
LEUKOPENIA (Blood and lymphatic system disorders) | 16 (19) | 15 (20) | 8 (10) | 4 (4) | 1 (1) | 3 (8) | 21 (30) | 10 (14) | 9 (15) | 10 (16) | 4 (5) | 20 (23)
LYMPHOPENIA (Blood and lymphatic system disorders) | 10 (15) | 15 (17) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 13 (26) | 6 (9) | 1 (2) | 10 (12) | 6 (6) | 17 (24)
NEUTROPENIA (Blood and lymphatic system disorders) | 11 (11) | 21 (28) | 16 (20) | 1 (1) | 3 (3) | 3 (3) | 14 (26) | 14 (16) | 17 (26) | 8 (11) | 7 (10) | 12 (18)
DIARRHOEA (Gastrointestinal disorders) | 23 (25) | 23 (26) | 19 (20) | 10 (10) | 5 (5) | 4 (4) | 14 (14) | 9 (9) | 10 (10) | 7 (7) | 8 (8) | 7 (9)
PYREXIA (General disorders) | 2 (4) | 16 (19) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 8 (9) | 5 (5) | 3 (3) | 9 (10) | 6 (7) | 8 (10)
BRONCHITIS (Infections and infestations) | 28 (30) | 33 (39) | 13 (14) | 10 (10) | 6 (6) | 3 (3) | 27 (33) | 12 (15) | 16 (18) | 16 (19) | 6 (6) | 25 (32)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 132 (150) | 51 (52) | 106 (119) | 57 (67) | 29 (30) | 117 (132)
HERPES ZOSTER (Infections and infestations) | 10 (10) | 16 (17) | 2 (2) | 3 (3) | 4 (4) | 10 (11) | 29 (30) | 21 (21) | 8 (8) | 12 (13) | 10 (10) | 9 (9)
LATENT TUBERCULOSIS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 22 (22) | 4 (4) | 19 (19) | 17 (17) | 8 (8) | 5 (5)
NASOPHARYNGITIS (Infections and infestations) | 36 (49) | 45 (52) | 43 (56) | 21 (24) | 7 (10) | 16 (18) | 38 (54) | 24 (27) | 31 (46) | 15 (22) | 9 (11) | 36 (46)
ORAL HERPES (Infections and infestations) | 11 (13) | 28 (43) | 10 (14) | 4 (4) | 2 (2) | 2 (2) | 9 (10) | 8 (19) | 9 (15) | 4 (5) | 5 (5) | 7 (10)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 67 (92) | 72 (100) | 53 (63) | 34 (37) | 13 (16) | 11 (13) | 56 (82) | 40 (52) | 42 (60) | 25 (48) | 15 (18) | 49 (62)
URINARY TRACT INFECTION (Infections and infestations) | 26 (37) | 30 (42) | 18 (21) | 10 (10) | 4 (6) | 9 (14) | 41 (64) | 21 (38) | 26 (32) | 15 (18) | 12 (18) | 25 (37)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 32 (45) | 39 (52) | 44 (53) | 12 (14) | 6 (6) | 8 (8) | 33 (48) | 23 (28) | 30 (35) | 18 (25) | 9 (15) | 19 (21)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 25 (29) | 29 (38) | 28 (32) | 8 (9) | 4 (4) | 9 (9) | 27 (38) | 23 (26) | 22 (28) | 14 (20) | 9 (12) | 18 (20)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 52 (69) | 67 (95) | 31 (38) | 6 (7) | 11 (13) | 15 (17) | 43 (76) | 33 (43) | 21 (34) | 22 (33) | 25 (32) | 39 (46)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (6) | 4 (4) | 2 (2) | 2 (2) | 4 (4) | 24 (34) | 8 (8) | 22 (27) | 13 (18) | 5 (5) | 15 (18)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (8) | 13 (13) | 11 (13) | 7 (8) | 0 (0) | 3 (6) | 29 (29) | 8 (8) | 18 (20) | 3 (3) | 8 (8) | 11 (11)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 12 (14) | 7 (8) | 14 (17) | 10 (12) | 3 (3) | 7 (7)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 14 (16) | 21 (21) | 20 (22) | 13 (14) | 2 (2) | 5 (5) | 42 (61) | 20 (24) | 33 (46) | 15 (19) | 10 (12) | 33 (42)
HEADACHE (Nervous system disorders) | 23 (32) | 21 (28) | 23 (24) | 10 (10) | 3 (6) | 2 (2) | 15 (42) | 13 (16) | 17 (20) | 6 (24) | 3 (3) | 12 (12)
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 23 (28) | 9 (9) | 5 (5) | 3 (3) | 3 (3) | 16 (17) | 7 (9) | 9 (12) | 9 (10) | 4 (4) | 13 (13)
PSORIASIS (Skin and subcutaneous tissue disorders) | 9 (10) | 8 (11) | 18 (20) | 8 (8) | 0 (0) | 0 (0) | 22 (24) | 20 (28) | 23 (29) | 12 (14) | 4 (4) | 26 (31)
HYPERTENSION (Vascular disorders) | 33 (37) | 21 (22) | 15 (15) | 10 (10) | 2 (2) | 2 (2) | 39 (44) | 11 (12) | 26 (27) | 15 (18) | 10 (10) | 20 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT03104400/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03104400/SAP_003.pdf